CLINICAL TRIAL: NCT03215212
Title: A Comparative Study to Assess the Effectiveness of Ear Plug, Eye Mask and Ocean Sound on Sleep Quality Among ICU Patients
Brief Title: Effectiveness of Ear Plug, Eye Mask and Ocean Sound on Sleep Quality Among ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Abhilasha Chaudhary, Student, M.sc Nursing, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 770
Record Dates: First submitted 2017-07-11; First posted 2017-07-12 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Sleep Quality
Keywords: ear plug; eye mask; ocean sound; sleep quality; intensive care unit
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Ear Protective Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- earplug (Experimental): Ear plug made from polyurethane with (NRR= 29 db and SNR= 37 db) administered from 10 pm to 7 am.
  Interventions: Other: eye mask; Other: ocean sound; Other: ear plug
- eye mask (Experimental): eye mask (18.5 cm, width 8.5cm, height -30mm )dark coloured cloth with 2 elasticised strap, covering both eyes administered from 10 pm to 7 am.
  Interventions: Other: eye mask; Other: ocean sound; Other: ear plug
- ocean sound (Experimental): Ocean sound a type of white noise administered via ear phone for 30 minutes from 9:15 pm to 9:45 pm
  Interventions: Other: eye mask; Other: ocean sound; Other: ear plug

INTERVENTIONS:
Other: eye mask — eye mask administered from 10 pm to 7 am
Other: ocean sound — Ocean sound administered via ear phone for 30 minutes from 9:15 pm to 9:45 pm
Other: ear plug — ear plug administered from 10 pm to 7 am

SUMMARY:
The study evaluates the effectiveness of ear plug, eye mask and ocean sound on sleep quality among ICU patients. 60 patients were randomly allocated to group 1 and group 2 by lottery method i.e 30 in each group. Group 1 received earplugs and eye masks on the first night followed by washout period on second night and received ocean sound on third night, while the group 2 received ocean sound on the first night followed by washout period on second night and received earplugs and eye mask on third night.

DETAILED DESCRIPTION:
a comparative study was done to assess the effectiveness of ear plug, eye mask and ocean sound on sleep quality.

Ear plug used in this study is a foam earplug made from polyurethane with noise reduction rating (NRR=29 dB, SNR=37dB). It is inserted into the ear canal to protect the user's ear from loud noise. The earplug used was manufactured by 3 M occupational health and environmental safety division company of India manufactured in Bengalaru560.Ear plug helps to reduce noise intensity which helps to decrease auditory perceptual processing.

Eye mask used in this study is a delicate dark colored cloth (black and blue) of fabric material, length -18.5 cm, width- 8.5cm, height- 30 millimeter filled with soft cushions like substance inside which cover both eyes and 2 elasticized strap that holds the mask on patients head which prevents incoming light away from patient's eyes and induces a state of pure darkness. The product detail of Eye mask was, model number-SM004 and was ordered from Amazon.Eye mask decreases the intensity of the light which enhances melatonin secretion (involve endocrine system). Additionally, eye mask helps to use of cognator subsystem as eye mask also helps to reduce visual perceptual processing.

Ocean sound is a type of white noise which is a soothing sound of waves crashing on the beach which is provided via ear phone for 30 min. It was delivered via the android application name relax melodies meditation of Ipnos software. Ocean sound is a type of white noise which prevents intense auditory stimuli less capable of stimulating the cerebral cortex during sleep which helps to decrease auditory perceptual processing.

ELIGIBILITY:
Inclusion Criteria:

* The patients who are 18 or more than 18 years of age.
* Patients who were oriented to the time and individual.
* Patients who could understand and respond in Hindi/English.
* Patients having no history of head trauma.
* Patients having no mental diseases.

Exclusion Criteria:

* Patients having any trauma in head, ears, and eyes.
* Patients reporting discomfort with eye mask and ear plug.
* Patients who had a hearing deficit.
* Patients taking sleep inducing drugs like Narcotics, Sedatives.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
sleep quality | 10-15 minutes
  structured sleep quality scale Scores for each question ranges from 0 to 3, with higher scores indicating poor sleep quality and lower score indicating good sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: abhilasha chaudhary, M.Sc Nursing, Principal Investigator — Maharishi Markandeshwar University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel M, Chipman J, Carlin BW, Shade D. Sleep in the intensive care unit setting. Crit Care Nurs Q. 2008 Oct-Dec;31(4):309-18; quiz 319-20. doi: 10.1097/01.CNQ.0000336816.89300.41. PMID 18815477
- [Background] Spencer JA, Moran DJ, Lee A, Talbert D. White noise and sleep induction. Arch Dis Child. 1990 Jan;65(1):135-7. doi: 10.1136/adc.65.1.135. PMID 2405784
- [Background] Wallace CJ, Robins J, Alvord LS, Walker JM. The effect of earplugs on sleep measures during exposure to simulated intensive care unit noise. Am J Crit Care. 1999 Jul;8(4):210-9. PMID 10392220
- [Result] Daneshmandi M, Neiseh F, SadeghiShermeh M, Ebadi A. Effect of eye mask on sleep quality in patients with acute coronary syndrome. J Caring Sci. 2012 Aug 25;1(3):135-43. doi: 10.5681/jcs.2012.020. eCollection 2012 Sep. PMID 25276688
- [Derived] Chaudhary A, Kumari V, Neetu N. Sleep Promotion among Critically Ill Patients: Earplugs/Eye Mask versus Ocean Sound-A Randomized Controlled Trial Study. Crit Care Res Pract. 2020 Dec 23;2020:8898172. doi: 10.1155/2020/8898172. eCollection 2020. PMID 33425385